CLINICAL TRIAL: NCT06299891
Title: Phentermine/Topiramate in Children, Adolescents, and Young Adults With Hypothalamic Obesity: a Pilot and Feasibility Study
Brief Title: Efficacy and Safety of Phentermine/Topiramate in Youth With Hypothalamic Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Christian L Roth, MD, Principal investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PhT_HypOb_Protocol_Clean_07-05
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hypothalamic Obesity; Hypothalamic Tumor; Craniopharyngioma
Keywords: Hypothalamic Lesion; Drug Intervention; Hypothalamic Obesity; Phentermine/Topiramate
MeSH Terms: conditions — Sexual Infantilism; Hypothalamic Neoplasms; Craniopharyngioma | interventions — Phentermine; Qsymia

STUDY DESIGN:
Intervention Model Description: Two-center, double-blind (participant and assessor), randomized, parallel-arm placebo-controlled 28-week clinical trial, comparing changes related to active drug (Qsymia®) vs. placebo (matched capsules).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible subjects will be assigned treatment using a sex-stratified permuted-block randomization (1:1) to drug vs. placebo for 28 weeks with varying block sizes constructed by the study statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug Intervention (Experimental): Active drug dose escalation and adjustment: The drug had been used in adolescents with obesity before. For this trial, the FDA approved dose titration will be followed until the highest tolerable dose is reached.
  Interventions: Drug: Phentermine / Topiramate Extended Release Oral Capsule [Qsymia]
- Placebo (Placebo Comparator): Matching placebo using capsules matching the appearance of the active drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Phentermine / Topiramate Extended Release Oral Capsule [Qsymia] — To assess safety and maximum tolerated dose as well as efficacy on weight loss of Phentermine/Topiramate in individuals with hypothalamic obesity.
  Arms: Drug Intervention
Other: Placebo — To assess safety and maximum tolerated dose as well as efficacy on weight loss of placebo treatment in individuals with hypothalamic obesity.
  Other Names: Matching blinded placebo capsules
  Arms: Placebo

SUMMARY:
Hypothalamic obesity (HO) refers to the substantial weight gain that often complicates hypothalamic brain tumors. Children with this treatment-recalcitrant form of obesity have excess rates of metabolic sequelae compared to otherwise healthy children with similar obesity, and later experience excess mortality related to cardiometabolic disease. In this pilot trial, our objective is to gather key preliminary data about phentermine/topiramate (Ph/T) that is FDA-approved for "common" obesity but has never been tested in HO. The subset of individuals with HO who experience hyperphagia or excess daytime sleepiness may benefit from the Ph/T-induced decrease in appetite and increase in alertness.

Preliminary assessments of safety, adverse events, dosing (Aim 1), as well as of efficacy (% BMI loss, Aim 2) will be made in a 28-week parallel-arm double-blinded Phase 2 placebo-controlled clinical trial in 6-28-year-old individuals with HO.

DETAILED DESCRIPTION:
STUDY OVERVIEW This is a two-center, double-blind (participant and assessor), randomized, parallel-arm 28-week clinical phase II trial, comparing changes from pre- to post treatment in two study arms of active drug (Qsymia®) vs. placebo capsules. Twenty-four 6-28-year-old participants will be randomized 1:1 into the two intervention groups. The study will have a single central IRB (CHOP).

In this pilot trial, the objective is to gather key preliminary data about phentermine/topiramate (Ph/T), a promising option containing a sympathomimetic amine (Ph) combined with an appetite-suppressive epilepsy drug (T) that is FDA-approved for "common" obesity but has never been tested in HO. The subset of individuals with HO who experience hyperphagia or excess daytime sleepiness may benefit from the Ph/T-induced decrease in appetite and increase in alertness. Preliminary assessments of safety and dosing (adverse events and maximum tolerated dose - Aim 1), as well as of efficacy (% BMI loss - Aim 2) will be made in a 28-week parallel-arm double-blinded Phase 2 randomized placebo-controlled clinical trial in 6-28-year-old individuals with HO. The FDA-approved dose titration will be followed. Other efficacy and mechanistic outcomes will be measured as well.

Specific Aims:

Aim 1: To assess safety and maximum tolerated dose of Ph/T. Main outcomes: treatment-emergent adverse events (including any during withdrawal), maximum tolerated dose (weeks 0 to 28).

Aim 2: To estimate the treatment effect of Ph/T with respect to weight loss in individuals with HO. Main outcome: % change in BMI (week 0 to 28) in response to Ph/T vs. placebo.

Study Approach:

Recruitment. Subjects will be required to travel to one of the two research sites (Seattle WA; Philadelphia PA). Each subject will be treated for 28 weeks plus 1 week of an appropriate taper in those participants who reached the highest dose at titration.

Participants will be pre-screened for eligibility via medical record review. Once written informed consent is obtained, eligibility will be confirmed.

Randomization. Eligible subjects will be assigned treatment using a permuted-block randomization (1:1) to drug vs. placebo for 28 weeks with varying block sizes constructed by the CHOP study statistician.

Study visits. Each participant will have a screening visit and 5 in-person study visits: Weeks 1 (baseline), 3, 14, 16, 28 (end of randomized trial). There will be a remote contact one week (+/- 3 days) after dose initiation and/or dose escalation to assess dose tolerability. The remote contact at 29 weeks will be performed to assess for any withdrawal effects and will be done in-person if there are any safety concerns that are most appropriately assessed in person. Visits at 1 and 28 weeks will be used for main outcome collection. Interim visits are required for assessment of dose escalation. Weeks 3 and 16 visits could be done remotely to reduce burden, in particular for individuals traveling from a distance, if participants prefer and have no concerning safety signals. Participants will be compensated for their time and travel. Efforts will be made to schedule study appointments at times that will accommodate participants' schedules.

Main outcome for Aim 1: Safety, as assessed by systematic collection of treatment-emergent adverse events using a safety monitoring uniform report form (SMURF), with adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

Secondary outcome for Aim 1: Maximum tolerated dose of Ph/T, as defined by the dose of Ph/T that the participant is continuing to take at the week 28 visit, reflecting any dose individualization.

Main outcome for Aim 2: % change in BMI between weeks 1 (baseline) and week 28 (end of treatment).

Key secondary outcomes for Aim 2 (all assessed as change between weeks 1 and 28): proportion of participants who achieve at least 2.5% BMI reduction, proportion of participants who achieve at least 5% BMI reduction, change in fat mass and visceral fat (as assessed by DXA) from Baseline to Week 28.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females; Ages 6-28 years (inclusive)
2. History of rapid weight gain related to tumor onset or treatment, as assessed by an experienced endocrinologist (for example, change in BMI z-score > 0.2 and/or BMI +5% during the first 6 months following tumor treatment)
3. Obesity (BMI > 95th%ile for age/sex using CDC 2000 reference for under 18; BMI > 30 kg/m2 for 18+ years)
4. Recent evidence of hypothalamic injury by brain MRI with central review; >6 months status-post definitive therapy (surgery, chemotherapy, or radiation); no major operations/surgeries planned during the study period.
5. Stable on pituitary replacement* and/or appetite-modulating medications (including stimulants) for at least 2 months. *Adjustments of less than 25% (<25%) are permitted to hydrocortisone, growth hormone or thyroid hormone. Sex steroids and DDAVP are exempt.
6. Post-menarchal females must use a highly effective form of contraception, unless hypogonadotropic hypogonadism is documented. All participating females of child-bearing potential will have pregnancy testing as outlined in the protocol.
7. Participants must be able to communicate well with the investigative team, must comply with requirements of the study, and be able to provide written informed consent and/or assent for individuals less than 18y with consent of a parent/legal guardian.

Exclusion Criteria:

1. Contraindication to Phentermine, Topiramate, or Qsymia as assessed using current package inserts. Including: History of glaucoma and known hyperthyroidism.
2. Known history of nephrolithiasis (kidney stones).
3. Current clinical diagnosis of anorexia nervosa or bulimia nervosa in the medical record.
4. Known history of metabolic acidosis, low bicarbonate on screening laboratory assessment (below lower limit of normal), or clinically significant bone disease requiring medication (beyond calcium and/or vitamin D).
5. Current or recent (<14 days) use of monoamine oxidase inhibitor.
6. Known hypersensitivity to sympathomimetic amines.
7. Clinically significant cardiovascular conditions, as defined as any of the following: i) abnormal blood pressure, defined as: under 13y, 95th%ile +12 mm Hg or > 140/90, whichever is lower; 13y and older, > 140/90 ; ii) history of cardiac arrhythmia or arrhythmia detected on screening ECG; iii) history of heart failure and/or cardiomyopathy; iv) prolonged QTc interval (QTc > 460 msec), and/or long QT syndrome phenotype and/or positive genotype for long QT syndrome pathogenic; v) history of cardiac disease including coronary artery disease.
8. Females who are pregnant, breastfeeding, or planning to become pregnant during the trial.
9. "Brittle" diabetes insipidus (in the opinion of the referring endocrinologist, e.g. requiring frequent hospitalizations and/or frequent abnormal sodium values).
10. Diabetes mellitus requiring insulin/secretagogue. HbA1c > 8.5% at Screening.
11. Clinically significant hyperthyroidism as assessed using thyroid hormone measurements. Clinical measurements within 12 months of baseline/screening may be used to assess this criterion.
12. History of clinically significant hypokalemia (low potassium) or current clinically significant hypokalemia (low potassium) on baseline/screening labs.
13. Clinically significant liver disease and/or known severe hepatic impairment. ALT > 3 x Upper Limit of Normal (ULN) AST > 3 x ULN
14. Clinically significant kidney disease. GFR<60 ml/min/1.73m2
15. History of seizure in the 12 months prior to Screening.
16. History of substance abuse, depression of moderate or greater severity, psychiatric disorder and/or suicidality.
17. History of abdominal surgery including gastric bypass.
18. Current use of supra-physiologic steroids.
19. History of allergy or sensitivity to test agents. Including individuals with known aspirin allergy or hypersensitivity and/or known allergy to FD&C Yellow No. 5 (tartrazine).
20. Concurrent use of carbonic anhydrase inhibitors.
21. Concurrent use of non-potassium sparing diuretics.
22. New weight management medication (or >5% decrease in weight over prior 2 months on any current, stable regimen), stimulant, and/or investigational medication within 2 months prior to screening, and/or plans to initiate other new weight management regimen.
23. Cognitive impairment that, in the opinion of the investigator, precludes participation in the study.
24. Individuals considered, in the Investigator's opinion, not suitable to participate in the study for reasons other than those indicated above.

Ages: 6 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | From baseline to completion of week 28
  Incidence of treatment-emergent adverse events including any during withdrawal in study drug vs. placebo.

SECONDARY OUTCOMES:
Maximum tolerated dose | Week 0 to 28
  Maximum tolerated dose achieved by the end of the study in study drug vs. placebo.
% change in BMI | Week 0 to 28
  % change in BMI in response to study drug vs. placebo.
Proportion of individuals who experience 5% decrease in BMI | Week 0 to 28
  Proportion of individuals who experience 5% decrease in BMI in response to study drug vs. placebo.
Proportion of individuals who experience 2.5% decrease in BMI | Week 0 to 28
  Proportion of individuals who experience 2.5% decrease in BMI in response to study drug vs. placebo
Change in body fat mass | Week 0 to 28
  Change in body fat mass via DXA in response to study drug vs. placebo.
Change in visceral fat mass | Week 0 to 28
  Change of visceral fat mass in response to study drug vs. placebo via DXA.
Change in hunger | Week 0 to 28
  Daily assessment of hunger by questionnaire scores will be recorded prior to the patient's first meal of the day.
Change in energy intake | Week 0 to 28
  Patient's dietary intake via the Automated Self-Administered 24-Hour Dietary Recall.

CONTACTS AND LOCATIONS:
Overall Officials: Christian L Roth, MD, Principal Investigator — University of Washington, Dept. of Pediatrics; Shana E McCormack, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No